CLINICAL TRIAL: NCT02115399
Title: ADRN Barrier/Immunoprofiling Exploratory Pilot Study (ADRN-04)
Brief Title: ADRN Barrier/Immunoprofiling Exploratory Pilot Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT ADRN-04
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Dermatitis; Dermatitis, Atopic; Eczema; Non-atopic Healthy Controls
Keywords: Dermatitis; Staphylococcus; Staphylococcus aureus; Dermatitis, Atopic; Non-atopic controls
MeSH Terms: conditions — Dermatitis; Dermatitis, Atopic; Eczema; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, skin tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ADStaph-: Atopic Dermatitis without a history of Eczema Herpeticum and without S. aureus skin colonization. A minimum of 45 participants will be enrolled in this group.
- ADStaph+: Atopic Dermatitis without a history of Eczema Herpeticum and with S. aureus skin colonization. A minimum of 45 participants will be enrolled in this group.
- NAStaph-: Non-atopic healthy participants without S. aureus skin colonization. A minimum of 45 participants will be enrolled in this group
- NAStaph+: Non-atopic healthy participants with S. aureus skin colonization. As the NAStaph+ phenotype is expected to be rare, as many participants as possible will be enrolled in this group; however, we do not expect to enroll 45 participants in this group.

SUMMARY:
The purpose of this study is to look at how defects in the skin barrier and immune response affect risk for skin infections.

Participants will be classified into 4 groups based on Atopic Dermatitis (AD)/Non-Atopic (NA) status and Staphylococcus aureus (S. aureus) colonization (negative or positive):

* AD S. aureus negative
* AD S. aureus positive
* NA S. aureus negative and
* NA S. aureus positive.

DETAILED DESCRIPTION:
Atopic dermatitis, also called eczema, is a disease in which the skin is dry and scaly with severe itching. People with atopic dermatitis have defects in the skin barrier as well as defects in the immune system which fights off skin infections. People who have atopic dermatitis often have complications from viral and bacterial skin infections, such as recurring Staphylococcus aureus (S. aureus), or Staph infections.

The study will compare the skin barrier and immune response of people with and without atopic dermatitis in relation to whether Staph bacteria is growing on their skin.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling all of the following criteria are eligible for enrollment-

* Non-Hispanic Caucasian males and females 18 to 60 years of age, inclusive, at the time of Enrollment
* Who are enrolled in the ADRN Registry study
* Who have active AD (lesions present) with or without a history of Eczema Herpeticum (EH) as defined in the ADRN Standard Diagnostic Criteria OR who meet criteria for the NA diagnostic group as defined in the ADRN Standard Diagnostic Criteria
* Who are willing to sign the informed consent form prior to initiation of any study procedures.

Exclusion Criteria:

Participants fulfilling any of the following criteria are not eligible for enrollment-

* Who are pregnant
* Who have an active systemic malignancy. Uncomplicated non-melanoma skin cancer and melanoma in situ with documentation of complete excision are not exclusionary
* Who have any skin disease other than AD that might compromise the SC barrier (e.g., bullous disease, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease)
* Who have a history of systemic immunological illness (e.g., human immunodeficiency virus [HIV] or systemic lupus erythematosus [SLE]) other than the condition being studied
* Who have active EH or eczema vaccinatum (EV)
* Who have a history of serious or life-threatening reaction to latex, tape, or adhesives
* Who are determined to be not eligible based on the opinion of the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants enrolled in the ADRN Registry study (NCT01494142) who fulfill eligibility criteria for this (ADRN04) study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The area under the transepidermal water loss (TEWL) curve | 6 month
  TEWL will be assessed using the AquaFlux AF200 (Biox, London UK) Transepidermal water loss (TEWL) will be assessed on non-lesional skin prior to tape stripping and repeated after 5, 10, 15, and 20 tape strips

SECONDARY OUTCOMES:
Basal transepidermal water loss (TEWL) | 6 month
  TEWL will be assessed using the AquaFlux AF200 (Biox, London UK)
Transepidermal water loss (TEWL) measured after 20 tape strips | 6 month
  Transepidermal water loss (TEWL) will be assessed using the AquaFlux AF200 (Biox, London UK). TEWL assessments will be done on non-lesional skin prior to tape stripping and after 20 tape strips and on unstripped lesional skin.
Change in transepidermal water loss (TEWL) | 6 month
  Transepidermal water loss (TEWL) will be assessed using the AquaFlux AF200 (Biox, London UK).
  TEWL after 20 tape strips minus transepidermal water loss (TEWL) prior to tape stripping.
Change in transepidermal water loss (TEWL) per every 5 tape strips (i.e. slope) | 6 month
  TEWL will be assessed using the AquaFlux AF200 (Biox, London UK)
Stratum Corneum (SC) hydration (capacitance) | 6 month
  Stratum Corneum(SC) hydration will be assessed on lesional and non-lesional skin using the Corneometer® CM825
Surface pH | 6 month
  Surface pH will be assessed on lesional and non-lesional skin using the Skin-pH Meter® PH 905
Stratum Corneum (SC) cohesion assessed as total protein removed per D-Squame tape | 6 month
  The assessment of SC cohesion will be conducted by two different methods. First, serial measurements of transepidermal water loss (TEWL) will be performed after tape stripping. Second, the amount of protein removed per strip will be calculated by an optical absorbance technique using a CuDerm SquameScan 850A.
Peripheral blood mononuclear cells (PBMC) expression of cell surface and intracellular markers | 6 month
  Measured after ex vivo stimulation with a polyclonal T cell stimulus, toll-like receptor ligands (TLRs), iron-regulated surface determinant B (IsdB) as an immunodominant S. aureus antigen, and recall antigens, such as influenza and tetanus antigens, and media alone as the control.
Itch assessment | 6 month
  Standardized questionnaires will be used to collect information regarding contact itch intensity
Quality of Life (QoL) measurement | 6 month
  Standardized questionnaires will be used to collect information regarding Quality of Life
Transepithelial Electrical Resistance (TEER) assessment from skin biopsies | 6 month
  Two punch biopsies of non-lesional skin will be obtained. One biopsy will be used for assessments of Tight Junction (TJ) function including confocal imaging, Transepithelial Electrical Resistance (TEER), and permeability measurements
Permeability assessment from skin biopsies | 6 month
  Two punch biopsies of non-lesional skin will be obtained. One biopsy will be used for assessments of Tight Junction (TJ) function including confocal imaging, Transepithelial Electrical Resistance (TEER), and permeability measurements.
Confocal staining of Tight Junction (TJs) from skin biopsies | 6 month
  Two punch biopsies of non-lesional skin will be obtained. One biopsy will be used for confocal staining of Tight Junction (TJs) and routine histology.
Atopic Dermatitis (AD) severity assessments | 6 month
  AD severity assessments include the Eczema Area and Severity Index (EASI), Rajka-Langeland (R-L) score, and Investigator Global Assessment (IGA)
Analysis of S. aureus isolates for antibiotic sensitivity | 6 month
  Antibiotic resistance is characterized by methicillin sensitive Staphylococcus aureus (MSSA) vs. methicillin resistant Staphylococcus aureus (MRSA)
Analysis of S. aureus isolates for expression of virulence or other factors | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Beck, MD, Study Chair — University of Rochester
Locations (3):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - University of Rochester, Rochester, New York
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/